CLINICAL TRIAL: NCT03916705
Title: Thoraco-Lumbar Fascia Mobility in Persons With Chronic Low Back Pain
Brief Title: Thoraco-Lumbar Fascia Mobility
Acronym: TLFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TLFM
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain
Keywords: Back Pain; Ultrasound; Fascia
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: Proof of concept study evaluating potential mechanisms of high-velocity low-amplitude spinal manipulation
Masking Description: Data analysis will be performed by blinded personnel. As a single group trial involving a manual therapy, participant and provider blinding is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single study arm (Other): All enrolled participants will undergo ultrasound evaluation and chiropractic low back spinal manipulation treatment.
  Interventions: Other: High Velocity Low amplitude spinal manipulation (HVLA-SM)

INTERVENTIONS:
Other: High Velocity Low amplitude spinal manipulation (HVLA-SM) — HVLA-SM is a commonly used spinal manipulation treatment for patients with chronic low back pain.

SUMMARY:
The purpose of the Thoraco-Lumbar Fascial Mobility (TLFM) study is to use ultrasound to measure the movement of connective tissue in the low back area of individuals with chronic low back pain (lasting more than 1 year). This study will compare baseline measurements, measurements after a single high velocity low amplitude spinal manipulation (HVLA-SM) and after a course of up to 16 HVLA-SM.

DETAILED DESCRIPTION:
The investigators will conduct a single arm pilot (proof-of-concept) clinical trial. Approximately 30 participants with self-reported chronic low-back pain (LBP), defined as pain for ≥ 1-year in duration and pain on at least ½ of the days in the past 6-months, will be enrolled.

This trial will consist of two separate enrollment phases. Phase 1 consists of enrollment at baseline followed by 3 separate ultrasound measurements. Phase 1 ends after a 4-week no treatment run-in phase.

Phase 2 begins twice-weekly HVLA-SM treatments to the thoracolumbar region for 8-weeks. Two ultrasound imaging evaluations will occur at visit 1 (pre and post-treatment). Pre-treatment ultrasound evaluations will be obtained at 4-weeks and 8-weeks.

The primary outcome is shear strain (adjacent tissue layer mobility measured with ultrasound) at the level of the lumbar L2-L3 vertebrae bilaterally. Ultrasound measures will be obtained with a Terason t3000 system using a 12L5 linear array probe with 10 MHz setting. Because shear strain may differ between sexes, we will attempt to recruit equal numbers of male and female participants.

ELIGIBILITY:
Inclusion:

1. Adults between 21 and 65 years
2. LBP of ≥ 1-yr duration with at least ½ of days with pain over the prior 6-months
3. Able to understand study procedures and willing to sign informed consent document
4. Willing to forgo any manual therapy for LBP for the initial 4-week study period
5. Willing to forgo any manual therapy for LBP other than study treatments during the 8-week treatment period
6. Able to tolerate and safely receive study procedures

Exclusion Criteria:

1. Chiropractic care or other manual therapy for at least 90 days prior to baseline visit
2. Unable to visualize necessary tissue layers using musculoskeletal ultrasound
3. Weight above 350 lbs
4. Unable to tolerate or safely receive study procedures
5. Need for referral
6. Unable or unwilling to comply with study procedures
7. Current or planned pregnancy (self-reported) within the study timeframe
8. Any prior surgery to the thoracolumbar region
9. Needing a proxy
10. Connective tissue disorder such as Marfan and Ehlers-Danlos syndrome

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Examine changes in thoracolumbar fascia movement (called shear-strain) using ultrasound | Short term change (Baseline), longer-term change (4 weeks)
  Short and longer-term changes in shear-strain will be studied by comparing between ultrasound recordings obtained at baseline and between measurements obtained at baseline and after 4-weeks
Investigate changes in thoracolumbar fascia movement (called shear-strain) using ultrasound after high-velocity low-amplitude spinal manipulation | 4-weeks, 8-weeks, 12 weeks
  Changes in shear-strain measures associated with high-velocity low-amplitude spinal manipulation will be assessed at 3 separate time points.
Examine differences in thoracolumbar movement (called shear-strain) using ultrasound. Measurements will be obtained in relaxed and active muscle contraction states | Baseline
  Compare thoracolumbar shear strain during relaxed passive flexion with active paraspinal contraction during passive flexion.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Global Health questions on pain intensity | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Worst, average, and current pain intensity measured on a self-reported 5-point numerical rating scale. Lower scores indicate lower pain
Patient Reported Outcomes Measurement Information System (PROMIS) Global Health questions of pain interference | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Pain interference measured on a self-reported 4-point numerical rating scale. The scale ranges from 4-20. Lower scores indicate higher pain interference.
Roland Morris Disability Questionnaire (RMDQ) | Baseline, 4 weeks, 8 weeks, and 12 weeks
  A 24-item self-reported scale assessing low-back pain related disability. Scores range from 0-24 with higher scores indicating higher disability.
Patient Reported Outcomes Measurement Information System (PROMIS) nociceptive pain quality scale | Baseline
  A 5-item self-reported scale used to identify persons more likely to have nociceptive pain. The scale ranges from 5-25 with higher scores indicating nociceptive pain is more likely.
Perceived Global Low Back Pain Improvement | 12 weeks
  A single question asking patients about their perceived improvement on a 7 point scale. Lower scores indicate greater improvement.
Patient Reported Outcomes Measurement Information System (PROMIS) neuropathic pain quality scale | Baseline
  A 5-item self-reported scale used to identify persons more likely to have neuropathic pain. The scale ranges from 5-25 with higher scores indicating neuropathic pain is more likely.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vinining, DC, DHSc, Principal Investigator — Palmer College of Chiropractic
Locations (1):
- Palmer Center for Chiropractic Research, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
This is a proof of concept study. No data will be available for sharing.

REFERENCES:
- [Derived] Vining R, Onifer SM, Twist E, Ziegler AM, Corber L, Long CR. Thoracolumbar fascia mobility and chronic low back pain: Phase 1 of a pilot and feasibility study assessing repeated measures and the influence of paraspinal muscle contraction. J Bodyw Mov Ther. 2023 Apr;34:19-27. doi: 10.1016/j.jbmt.2023.04.004. Epub 2023 Apr 6. PMID 37301552
- [Derived] Vining R, Onifer SM, Twist E, Ziegler AM, Corber L, Long CR. Thoracolumbar fascia mobility and chronic low back pain: Phase 2 of a pilot and feasibility study including multimodal chiropractic care. Chiropr Man Therap. 2022 Oct 21;30(1):46. doi: 10.1186/s12998-022-00455-z. PMID 36271428

DOCUMENTS (1):
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03916705/ICF_000.pdf